CLINICAL TRIAL: NCT06390124
Title: Reconstructive Therapy of Advanced Peri-implantitis-related Bone Defect with PDGF-BB (Gem-21)
Brief Title: Reconstructive Therapy of Peri-implantitis with PDGF-BB (Gem-21)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Principal Investigator, Alberto Monje, Head of department of Periodontology, Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 311022
Record Dates: First submitted 2024-03-20; First posted 2024-04-30 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-04

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Platelet-Derived Growth Factor

STUDY DESIGN:
Intervention Model Description: Prospective case series
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental group (Experimental): Platelet derived growth factor (PDGF) is to be used to soak the implant surface and in combination with the bone grafting material
  Interventions: Drug: Platelet Derived Growth Factor (PDGF)

INTERVENTIONS:
Drug: Platelet Derived Growth Factor (PDGF) — Reconstructive therapy of advanced peri-implantitis-related defects with anorganic bovine bone and allograft combined with PDGF

SUMMARY:
Peri-implantitis is considered a bacteria-mediated inflammatory disease that leads to a progressive loss of support. During the last decade, research has been striving to understand this entity and strategies for primary and secondary prevention of the disease; However, all of them are about the effectiveness of different therapeutic modalities for their management. In general, it was stated that surgical therapy was ineffective in resolving inflammation. Therefore, surgical strategies are usually needed to eradicate the pathology.

Taking advantage of the knowledge acquired during approximately a period of time about the surgical treatment of periodontitis, if you propose several alternatives. These are mainly based on the morphology of the defect, although other factors, such as the lack of keratinized mucosa or the habit of smoking can alter the decision-making process. As such, peri-implantitis with angular defects (i.e., defects with infraosseous components) is indicated for reconstructive measurements with no barrier membranes. On the other hand, horizontal defects (i.e., defects with supra-crestal components) are more likely to resolve by resecting therapy with or without bone contouring measures.

It is interesting to note that, although early data indicated that the morphology of the peri-implantitis defect often shows a well-contained circumferential defect, it has recently been shown that it often presents a 2/3 wall defect configuration, where the buccal plate is commonly missing bone wall. The reason for this characteristic may recur in the dimension of the basal alveolar bones, insufficient critical buccal bone thickness or implant positioning13 in relation to the bone envelope. In addition, it should be noted that ~ 25% of peri-implantitis diagnosed on a daily basis exhibit a combined configuration of defects (i.e., a combination of infraosseous and supra-critical components).

For their reconstructive treatment, many biomaterials have been documented, among them several protocols proposed by our research group. However, the use of biological agents or growth factors has not been investigated for a long time. Platelet Derived Growth Factor (PDGF, Platelet Derived Growth Factor) is one of several Growth Factors or proteins that regulate cell growth and Cellular Division. PDGF plays a significant role, especially for Angiogenesis, which implies the growth of blood vessels from the existing vascular tissue. Uncontrolled angiogenesis is characteristic of cancer. Chemically the PDGF is a Glucoprotein chains A (-AA) or B (-BB) or composed of them (-AB). In the field of periodontics, periodontal regeneration has been shown to be successful in obtaining radiographic bone gain and tissue regeneration.

ELIGIBILITY:
All the sujects had dental implants with implant prostheses supported or removable or hardened for a minimum of 36 months. The following criteria should be applied: all patients aged 18 to 80 years, non-smokers, in the presence of systemic disease or medication that alters bone metabolism, and partial or complete edentulous patients who do not have active periodontal disease. The subjects were excluded due to: pregnancy or lactation, history or current smokers, uncontrolled medical conditions, case-hardened restorations, lack of keratinized mucosa (≤2 mm) at the sites of lingual or oral implantation and advanced peri-implantitis (A) (> 6 mm /> 50% of the implant length).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Rate of disease resolution | 12 months after surgery
  pockets <6mm with no bleeding on probing

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Monje, DDS, Principal Investigator — CICOM, Badajoz, Spain
Locations (1):
- Centro de Implantologia Cirugia Oral y Maxilofacial, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The goal is to publish the data in a scientific journal.